CLINICAL TRIAL: NCT06624566
Title: EINTER PROGRAM: Intensive Therapeutic Exercise in Patients With Spinal Cord Injury.
Brief Title: EINTER PROGRAM in Spinal Cord Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024.161
Record Dates: First submitted 2024-09-11; First posted 2024-10-03 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-09

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injuries; Physical Exercise; resistance; strength; exercise program
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: Study design Quasi-experimental single-group study with pre-post design. Participants:
  Inclusion/exclusion criteria o Inclusion criteria: adult patients with 18 years diagnosed with spinal cord injury below C3 admitted to the Neurorehabilitation ward of the Miguel Servet University Hospital.
  Exclusion criteria: Patients with tetraplegia with level C3.
Masking Description: As a quasi-experimental observational study, there is no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The A group received a program of therapeutic physical exercise scheduled from Monday to Friday (Experimental): The program protocol for group A consists of: Mondays and Wednesdays: Aerobic circuit protocol (45').
  * Warm-up 1-5 min: Global exercises, gentle stretching and range of motion exercises;
  * Aerobic exercise 30 min, at a target heart rate of 70% FCR in wheelchair. Aerobic exercises will consist of the use of different exercise programs using the "Motomed" type motorized kinesitherapy equipment.
  * Cool down 5-10 min. Tuesday and Thursday: Strength circuit protocol (45')
  * Warm up 1-5 min: global exercises, gentle stretching and range of motion exercises.
  Strength training 30 min:
  * Concentric and eccentric upper extremity muscle training. Also lower extremity muscle training (hip extensors/flexors and adductors/abductors, knee flexors and extensors, dorsal and plantar ankle flexors). 3 sets/10 repetitions for each exercise at 50-80% RM.
  * Cool down for 5-10 min.
  Friday: Combined workout (45'):
  * 20min aerobic protocol and 15 min strength protocol.
  * 5-10 min cool down.
  Interventions: Other: Experimental: Implementation of an intensive therapeutic group exercise program in the neurorehabilitation process
- The B group received a program of therapeutic physical exercise scheduled from Monday (Experimental): The program protocol for group B consists of: Monday and Wednesday: Aerobic circuit protocol (45'). o Warm-up 1-5 min: Global exercises, gentle stretching and range of motion exercises; aerobic exercises, consisting of graded walking, step or stationary bike, each at a target heart rate of 70% FCR. o Cool down 5-10 min. Tuesday and Thursday: Strength circuit protocol (45') o Warm up 1-5 min: global exercises, gentle stretching and range of motion exercises. o Strength training 30 min: Concentric and eccentric upper extremity muscle training. Also lower extremity muscle training (hip extensors/flexors and adductors/abductors, knee flexors and extensors, dorsal and plantar ankle flexors). 3 sets/10 repetitions for each exercise at 50-80% RM. Cool down for 5-10 min. Friday: Combined workout (45'): o 20min aerobic protocol and 15 min strength protocol. o 5-10 min cool down.
  Interventions: Other: Experimental: Implementation of an intensive therapeutic group exercise program in the neurorehabilitation process

INTERVENTIONS:
Other: Experimental: Implementation of an intensive therapeutic group exercise program in the neurorehabilitation process — Description: The variables will be measured prior to group assignment The age and sex variables and the satisfaction survey will be measured at the beginning of the program, the other variables at 20 sessions, at 40 sessions, at 60 sessions and/or at hospital discharge. Before the patient starts the program, he/she is classified in group A - patients who have seated trunk control for at least 2 minutes (with supervision) and no standing control (Berg scale item 3.3) - or in group B - patients who have standing trunk control for 2 minutes (with supervision) (Berg scale item 2.3). There is a maximum of 4 patients per group with 1 physiotherapist per group.. There is a maximum of 4 patients per group with 1 physiotherapist per group.. The difference with respect to the usual treatment of the neurorehabilitation service of the HMS is that in the EINTER program, strength and endurance exercises will be implemented in addition to the usual care plan

SUMMARY:
This study consists of the implementation of a therapeutic physical exercise program in a group setting in patients with spinal cord injury admitted to the Miguel Servet University Hospital in Zaragoza. This program consists of performing strength and endurance exercises from Monday to Friday with a duration of approximately 45 minutes each session.

The groups are created in such a way that the subjects in each group are homogeneous. This homogeneity is classified according to whether or not trunk control in seated or standing position is maintained in an autonomous manner as measured by the Berg scale. Each group consists of a maximum of 4 subjects and there are a maximum of 2 groups, and 1 physiotherapist per group. Group A is for those subjects who do not maintain independent standing, but maintain trunk control while seated, and group B is for those patients who do maintain independent standing.

Prior to the start of the program, subjects are informed of the study and evaluated with a series of health indicators (scales) to measure the impact of the program at the beginning of the program and at hospital discharge. These scales are as follows:

To measure muscular strength the investigators use the Medical Research Council, and to measure aerobic endurance the investigators use the 6 Minute Walking Test for patients who can ambulate autonomously and the 6 Minutes Pushing Test for those patients who do not ambulate and move around in a wheelchair. In addition, the investigators pass a satisfaction

DETAILED DESCRIPTION:
Metabolic alterations in patients with spinal cord injury are associated, among others, with arterial hypertension, lipid alterations, hyperinsulinemia and glucose transport disorders, which can lead to diabetes. This may favor the appearance of obesity phenomena in this type of patients. The decrease in physical exercise can increase these complications. With an increase in the level of physical activity, caloric expenditure is increased, thus improving the transport of glucose in the blood and decreasing the processes of diabetes. In addition, movement components such as strength and endurance are improved, which provides an improvement in balance. Therefore, with this increase in physical activity the investigators facilitate the patients greater participation in their environment once they are discharged from the hospital. Within the hospital setting, time away from scheduled therapy in patients with spinal cord injury on the Neurorehabilitation ward (U.L.M.E.) constitutes the majority of their waking time when they are admitted to this ward. Studies from other hospitals show that, as a rule, this time is approximately 4 hours a day, of which only 7-10 minutes a day are devoted to moderate and vigorous physical activity. For these reasons, the investigators consider it very important to implement therapeutic exercise programs in people with neurological pathology, in this case with a diagnosis of spinal cord injury, and to verify the impact it has on strength and endurance in this population.

The main hypothesis is that training through a designed program of therapeutic physical exercise optimizes the results referred to the improvement of strength and endurance in patients with spinal cord injury admitted to the Neurorehabilitation ward (U.L.M.E) of the Miguel Servet Hospital in Zaragoza.

The secondary hypotheses are that training based on a designed program of therapeutic physical exercise is satisfactory for patients with spinal cord injury admitted to the Neurorehabilitation ward of the Miguel Servet Hospital of Zaragoza.

The objectives of this study are:

1. To improve the strength of patients with spinal cord injury at the U.L.M.E.
2. To improve the aerobic endurance of the patient with spinal cord injury in the U.L.M.E.
3. To increase the patients adherence to physiotherapy treatments.
4. To assess patient satisfaction with their participation in therapeutic physical exercise programs.

Sources of information: Data regarding age, sex and metabolic variables are extracted from the electronic medical record. The strength and endurance variables are extracted from the assessment performed by the evaluating physiotherapists and saved in paper format and an Excel sheet. These variables are collected before starting the EINTER program and at hospital discharge. Likewise, at hospital discharge, a satisfaction survey and a personalized exercise sheet are provided. The variables collected are: o Muscular strength measured by the Medical Research Council o Aerobic endurance measured by the 6 Minute Walking Test for patients who can walk independently and the 6 Minutes Pushing Test for those patients who do not walk and move around in a wheelchair. o Adherence measured by the number of sessions in which the patient has participated o Satisfaction survey.

Before the patient starts the program, he/she is classified in group A -patients who have seated trunk control for at least 2 minutes (with supervision) and no standing control (Item 3.3, Berg scale)- or in group B -patients who have standing trunk control for 2 minutes (with supervision) (Item 2.3 on the Berg scale)-. There is a maximum of 4 patients per group with 1 physiotherapist per group.

Statistical analysis For statistical analysis the program R Ver. 4.1.3 (R Foundation for Statistical Computing, Institute for Statistics and Mathematics, Welthandelsplatz 1, 1020 Vienna, Austria) will be used. The significance level will be set at p&amp;amp;lt;0.05. The Kolmogorov-Smirnov test with Lilliefors correction will be used to test the distribution of quantitative variables. Quantitative variables will be described with mean±standard deviation or median [interquartile range] according to their distribution and qualitative variables with absolute and relative values (%). Pre-treatment differences will be analyzed with a t-test for related data or with the Wilcoxon signed-rank test for quantitative variables according to their distribution, and with Fishers exact text for qualitative variables. Limitations of the study One of the main limitations of the study is not being able to have a control group to be able to perform a Randomized Clinical Trial. Another limitation is the few variables incorporated in the study. For future studies, it would be interesting to introduce variables related to the social participation of the patient in his environment once discharged from hospital.

This study is based on an intervention based on therapeutic exercise, a tool that is within the scope of competence of physical therapists, therefore it is considered to be covered by the Civil Liability Insurance policy as professional members.

The project is planned to be carried out in the multifunctional room of the Neurorehabilitation Department of the Miguel Servet University Hospital of Zaragoza. The material to be used is the usual one for the professional practice of the physiotherapist and it is detailed below:

* 4 SETS OF DUMBBELLS OF DIFFERENT WEIGHTS
* 3 PULSE OXIMETERS
* 3 MEDICINE BALLS OF DIFFERENT WEIGHTS
* 3 PAIRS OF DIFFERENT WEIGHTS
* 1 STRETCHER
* 1 MOTOMED
* 1 PARALLEL BARS.

ELIGIBILITY:
Inclusion criteria:

Adult patients 18 years of age or older. Clinical diagnosis of spinal cord injury below C3 admitted to the Neurorehabilitation ward of the Miguel Servet University Hospital.

Exclusion criteria:

Clinical diagnosis of spinal cord injury level at C3 with tetraplegia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Strength | From the beginning of the program up to 12 weeks
  o Muscular strength measured by Medical Research Council
Resistance | From the beginning of the program up to 12 weeks
  o Aerobic endurance measured by the 6 Minute Walking Test for patients who can ambulate autonomously and the 6 Minutes Pushing Test for those patients who do not ambulate and move around in a wheelchair.

SECONDARY OUTCOMES:
Adherence to the program and level of satisfaction | From the beginning of the program up to 12 weeks
  Monitoring the number of sessions attended and by means of a satisfaction survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Miguel Servet, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No
Only numerical data of the primary and secondary variables, age and sex, totally anonymized, will be provided to the person responsible for the statistical analysis.

REFERENCES:
- [Result] Dupepe EB, Davis M, Elsayed GA, Agee B, Kirksey K, Gordon A, Pritchard PR. Inter-rater reliability of the modified Medical Research Council scale in patients with chronic incomplete spinal cord injury. J Neurosurg Spine. 2019 Jan 18;30(4):515-519. doi: 10.3171/2018.9.SPINE18508. Print 2019 Apr 1. PMID 30660112
- [Result] Solanki R, Chaudhari P, Bhise A. 60 :: Cardio Respiratory Fitness Testing in Spinal Cord Injury Patients Using 6 Minute Push Test Original Article Healthline Journal. 7(1).
- [Result] Martin Ginis KA, van der Scheer JW, Latimer-Cheung AE, Barrow A, Bourne C, Carruthers P, Bernardi M, Ditor DS, Gaudet S, de Groot S, Hayes KC, Hicks AL, Leicht CA, Lexell J, Macaluso S, Manns PJ, McBride CB, Noonan VK, Pomerleau P, Rimmer JH, Shaw RB, Smith B, Smith KM, Steeves JD, Tussler D, West CR, Wolfe DL, Goosey-Tolfrey VL. Evidence-based scientific exercise guidelines for adults with spinal cord injury: an update and a new guideline. Spinal Cord. 2018 Apr;56(4):308-321. doi: 10.1038/s41393-017-0017-3. Epub 2017 Oct 25. PMID 29070812
- [Result] Cowan RE, Callahan MK, Nash MS. The 6-min push test is reliable and predicts low fitness in spinal cord injury. Med Sci Sports Exerc. 2012 Oct;44(10):1993-2000. doi: 10.1249/MSS.0b013e31825cb3b6. PMID 22617394
- [Result] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Result] Hornby TG, Reisman DS, Ward IG, Scheets PL, Miller A, Haddad D, Fox EJ, Fritz NE, Hawkins K, Henderson CE, Hendron KL, Holleran CL, Lynskey JE, Walter A; and the Locomotor CPG Appraisal Team. Clinical Practice Guideline to Improve Locomotor Function Following Chronic Stroke, Incomplete Spinal Cord Injury, and Brain Injury. J Neurol Phys Ther. 2020 Jan;44(1):49-100. doi: 10.1097/NPT.0000000000000303. PMID 31834165
- [Result] Bauman WA, Spungen AM. Disorders of carbohydrate and lipid metabolism in veterans with paraplegia or quadriplegia: a model of premature aging. Metabolism. 1994 Jun;43(6):749-56. doi: 10.1016/0026-0495(94)90126-0. PMID 8201966